CLINICAL TRIAL: NCT06797154
Title: A Novel Wrist Wearable Sensor System to Promote Hemiparetic Upper Extremity Use in Home Daily Life of Subacute Stroke Survivors
Brief Title: A Novel Wrist Wearable Sensor System to Promote Hemiparetic Upper Extremity Use in Subacute Stroke Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: BioSensics (Industry); MGH Institute of Health Professions (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024P003622; R44HD084035 (NIH)
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Stroke Sequelae; Hemiparesis;Poststroke/CVA
Keywords: StrokeWear; Biosensics; Behavioral Intervention
MeSH Terms: conditions — Stroke | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- StrokeWear Motor and Behavioral Intervention (Experimental): Stroke survivors randomized to this group will receive standard rehabilitation (i.e., physical and occupational therapy) as well as a behavioral intervention aimed to encourage the use of the stroke affected arm during the performance of activities of daily living.
  Interventions: Behavioral: StrokeWear Behavioral Intervention
- Sham Comparator: Usual Care (Other): Stroke survivors randomized to this group will receive standard rehabilitation (i.e., physical and occupational therapy).
  Interventions: Other: Usual Care + Sham

INTERVENTIONS:
Behavioral: StrokeWear Behavioral Intervention — Behavioral strategies will be incorporated into the Strokewear system to encourage feedback on behavior, goal setting, daily activity action planning (DAAP), and an empowerment/ self management model to foster planned hemiparetic UE use during daily activities in the home and community. Patient empowerment in this study will occur over 6-months as patients gain the ability to use the StrokeWear technology independently and develop skills to self- manage their GDM and DAAP.
  Arms: StrokeWear Motor and Behavioral Intervention
Other: Usual Care + Sham — The intervention will consist in a sham version of the StrokeWear system and usual clinical care under the direction of a clinician. The sham version of the StrokeWear system will include sensing and recording technology to detect GDMs. However, study participants will not receive feedback from the system regarding the GDM counts.
  Arms: Sham Comparator: Usual Care

SUMMARY:
The proposed study is a two-arm randomized clinical trial designed to assess the effects of the StrokeWear system on clinical outcomes over a period of 6-months in subacute stroke survivors. The Intervention group will use StrokeWear system in combination to a motor and behavioral home intervention whereas the Control group will follow usual care which consists of a home-exercise plan (HEP).

DETAILED DESCRIPTION:
The proposed study is a two-arm randomized clinical trial designed to assess the effects of the StrokeWear system on clinical outcomes over a period of 6-months in subacute stroke survivors. The Intervention group will use StrokeWear system in combination to a motor and behavioral home intervention whereas the Control group will follow usual care which consists of a home-exercise plan (HEP).

Study participants will be asked to take part in 4 evaluation study visits: one screening and enrollment visit, and three evaluation visits (at baseline, at 3 months and at 6 months - at the intervention completion). Subject upper-extremity motor function will be assessed across domains of the International Classification of Functioning, Disability and Health (ICF) model. Groups will be stratified by baseline motor impairment and stroke chronicity.

Subjects randomized to the intervention group will take part of weekly coaching sessions during the first month, bi-weekly sessions during the months 2 and 3, and monthly sessions during months 4-6. These sessions will be held in-person or remotely, based on the study participant preference.

Subjects randomized to the control group will take part of monthly visits, held in-person or remotely (based on study participant preference), to re-evaluate the home-exercise plan and prescribe an update list of exercises for the following month.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-85 years of age at the time of enrollment
* Anterior circulation ischemic stroke at least 1 month and no more than 6 months prior to study enrollment;
* Unilateral upper extremity hemiparesis as characterized by initial scores on upper limb subtest of the Fugl-Meyer Assessment (FMA-UE) between 20 and 45;
* Intact cognitive function to understand the study procedures and goal setting (MMSE score above 23 and able to follow 3step command) ;
* Owning a smartphone (iOS or Android) and being familiar and comfortable with and owning a tablet or smartphone
* SAFE score equal or greater than 5

Exclusion Criteria:

* Severe spasticity (defined as a Modified Ashworth scale score of 3 or more) that would prevent safe performance of UE tasks;
* Visual impairments as assessed by the NIH Stroke Scale Visual Field subscale (only subjects with no visual loss will participate in the study); or hemispatial neglect that would impair the subject ability to see the feedback on the app screen (as assessed with the Mesulum cancellation test);
* Individuals with open wounds or recent fracture (less than 3 months) in the upper extremity, fragile skin or active infection;
* Upper-extremity orthopedic injuries or severe pain resulting in movement limitations;
* Diagnosis of other neurological disease; (i.e., Parkinson's disease, multiple sclerosis, ...);
* Severe proprioceptive deficits that impair the ability to process the vibration feedback, as assessed by physical examination during screening;
* Not understanding spoken or written English;
* Contralateral motor deficits as assessed by clinical examination;
* Brainstem and cerebellar stroke.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Motor Activity Log-Amount of Use | Change from baseline Motor Activity Log-Amount of Use score at 6 months
  Self-reported measure of upper-extremity performance. Score from 0 (worst) to 5 (best)
Change in Fugl-Meyer Upper-Extremity | Change from baseline Fugl-Meyer Upper-Extremity score at 6 months
  Observed measure of upper-extremity motor impairment following a stroke. Score from 0 (worst) to 66 (best)
Change in Upper-Extremity Activity Counts | Change from baseline Upper-Extremity Activity Counts score at 6 months
  Activity of the hemiparetic upper-extremity in the home setting as measured with wrist-worn accelerometers

SECONDARY OUTCOMES:
Change in Motor Activity Log-Quality of Use | Change from baseline Motor Activity Log-Quality of Use score at 6 months
  Self-reported measure of upper-extremity quality of use. Score from 0 (worst) to 5 (best)
Change in Wolf-Motor Function Test - Time subscale | Change from baseline Wolf-Motor Function Test - Time subscale score at 6 months
  Observed (timed) measure of upper-extremity function. Time from 0 to 120 seconds (maximum time allowed to attempt to perform a motor task)
Change in Wolf-Motor Function Test - Functional ability subscale | Change from baseline Wolf-Motor Function Test - Functional ability subscale score at 6 months
  Measure of upper-extremity quality of movement based on visual observation. Score from 0 (worst) to 5 (best)
Change in Stroke Impact Scale (SIS) | Change from baseline Stroke Impact Scale (SIS) score at 6 months
  Self-reported measure of quality of life after a stroke. Score from 0 (best) to 42 (worst)
Change in Stroke Self-Efficacy Questionnaire (SSEQ) - Activity subscale | Change from baseline Stroke Self-Efficacy Questionnaire (SSEQ) - Activity subscale score at 6 months
  Self-reported measure of upper-extremity efficacy in activities of daily living. Score from 0 (worst) to 10 (best).
Change in Stroke Self-Efficacy Questionnaire (SSEQ) - Self-management subscale | Change from baseline Self-Efficacy Questionnaire (SSEQ) - Self-management subscale score at 6 months
  Self-reported measure of upper-extremity efficacy in activities of daily living. Score from 0 (worst) to 10 (best).

OTHER OUTCOMES:
Number of times the activity goals are reached | At 6 months
  Number of times the activity goals set are reached over the study duration

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No